CLINICAL TRIAL: NCT01109017
Title: A Multicentre, Open Label, Observational, Non-interventional Study to Evaluate the Long-term Safety and Efficacy of Norditropin® Formulation in Patients With AGHD
Brief Title: Observational Study of the Safety and Efficacy of Norditropin® in Adult Patients With Growth Hormone Deficiency
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-3811; U1111-1114-6250 (Other: WHO); JapicCTI-101122 (Registry Identifier: JAPIC)
Record Dates: First submitted 2010-04-19; First posted 2010-04-22 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Norditropin®
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Norditropin® (somatropin) prescribed at the discretion of the physician according to normal clinical practice. Safety and effectiveness data is recorded by the physician, and a Quality of Life form is completed by the patient, at visits 1 to 5.

SUMMARY:
This study is conducted in Japan. The aim of this observational study is to collect information about the safety and efficacy of Norditropin® long-term treatment of growth hormone deficiency in adults.

ELIGIBILITY:
Inclusion Criteria:

* Severe adult growth hormone deficiency

Exclusion Criteria:

* Known or suspected allergy to study product(s) or related products
* Previous participation in the study
* Diabetes Mellitus
* Presence of malignant tumor(s)
* Pregnant or likely to get pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with growth hormone deficiency including newly-diagnosed patients, who are considered to need treatment with Norditropin® (somatropin) or already on therapy with Norditropin® (somatropin) are eligible for inclusion in the study
Sampling Method: Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2009-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number and type of suspected serious adverse drug reactions (SADRs) during the study period | after 5 years

SECONDARY OUTCOMES:
Number of impaired glucose tolerance events during the study period | evaluated after 3 months, 6 months, 1 year and between 2-5 years
Number of other types of adverse events (AEs) during the study period | evaluated after 3 months, 6 months, 1 year and between 2-5 years
Effects on body composition (body fat percentage, lean body weight mass, bone density, bone mineral density) | evaluated after 3 months, 6 months, 1 year and between 2-5 years
Effects of insulin-like growth factor-1 (IGF-I) levels | evaluated after 3 months, 6 months, 1 year and between 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com